CLINICAL TRIAL: NCT01077505
Title: An Open-label Study to Evaluate the Pharmacokinetics of an Oral Contraceptive Containing Norethindrone and Ethinyl Estradiol When Co-administered With GSK716155 in Healthy Adult Female Subjects
Brief Title: An Evaluation of the Pharmacokinetics of an Oral Contraceptive (Brevicon) When Co-administered With Albiglutide .
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 107032
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacokinetics; GSK716155; Brevicon; albiglutide; healthy female volunteers; oral contraceptive
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Contraceptives, Oral; norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- albiglutide (Experimental): albiglutide 50mg weekly
  Interventions: Biological: albiglutide; Drug: Oral contraceptive (Brevicon)

INTERVENTIONS:
Biological: albiglutide — albiglutide 50mg weekly subcutaneous injection
Drug: Oral contraceptive (Brevicon) — Oral contraceptive (Brevicon)

SUMMARY:
This study will be an open-label study to evaluate the effect of albiglutide on the pharmacokinetics and pharmacodynamics of a standard oral contraceptive regimen (Brevicon). The primary objective of this study is to demonstrate the lack of effect of albiglutide doses on the pharmacokinetics of norethindrone and ethinyl estradiol in healthy female subjects.

DETAILED DESCRIPTION:
This study will be an open-label study in at least one center to evaluate the effect of albiglutide administration on the pharmacokinetics and pharmacodynamics of a standard oral contraceptive regimen (Brevicon). The primary objective of this study is to demonstrate the lack of effect of albiglutide doses on the pharmacokinetics of norethindrone and ethinyl estradiol in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects, defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, clinical laboratory tests, and 12-lead ECG;
* Women of childbearing potential must use protocol-defined contraceptive methods;
* BMI is 19 to 30 kg/m2 and body weight ≥50 kg (110 lbs) and <114 kg (<250 lbs);
* Aspartate aminotransferase (AST), ALT, alkaline phosphatase, and bilirubin is </=1.5 × ULN;

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or ECG;
* Blood pressure ≥140/90 mm Hg or heart rate >100 beats/minute at Screening;
* Corrected QT (QTc) intervals >450 msec (per ECG machine interpretation);
* Pregnant or nursing females;
* A positive prestudy hepatitis B surface antigen, positive hepatitis C antibody, or HIV result within 3 months of Screening;
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
* Smoking or using any nicotine products, including smoking cessation patches containing any amount of nicotine within the 6 months before Screening;
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception;
* Subjects have participated in a clinical trial and have received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer);
* History of substance abuse within the past year as determined by the investigator;
* History of alcohol abuse defined as an average weekly intake of >7 drinks;
* Positive urine drug screen at Screening or predose during the Run-in Period and on Day 1 of Periods 1 and 2;
* Use of prescription or nonprescription drugs, vitamins, dietary/herbal supplements including St. John's Wort, nonsteroidal antiinflammatory medications, and aspirin within 14 days or 5 half-lives, whichever is longer prior to the first dose of investigational product;
* Willing to refrain from consuming grapefruit or cranberry products (such as juice, fruit, or nutritional supplements) at any time during participation in the study;
* Donation of blood in excess of 500 mL within 56 days prior to dosing or intention of donating in the month after completing the study;
* History of thyroid dysfunction or an abnormal (i.e., outside normal reference range) thyroid function test assessed by thyroid stimulating hormone (TSH) at Screening;
* History of drug allergy or other allergy, which, in the opinion of the responsible study physician, contradicts the subject's participation;
* History of any condition that would contraindicate OC administration (including hypertension, stroke, ischemic heart disease, venous thromboembolism, carcinoma of the breast, etc.);
* History of type 1 or 2 diabetes mellitus;
* History of migraine if aged >35 years or has focal symptoms associated with migraine;
* Any condition that would affect drug transit time or absorption (e.g., gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, chronic diarrhea, vagotomy, chronic gastroesophageal reflux disease, malabsorption, colostomy, Crohn's disease, ulcerative colitis, or celiac sprue); or
* Previous or current receipt of exenatide or any other GLP 1 agonist;

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03-15 (Actual); Primary Completion 2010-11-24 (Actual); Study Completion 2010-11-24 (Actual)

PRIMARY OUTCOMES:
AUC0-24 of norethindrone and ethinyl estradiol after OC alone in Period 1 and after OC with albiglutide in Period 2. | Day 21

SECONDARY OUTCOMES:
Cmax, Cmin, tmax, and t½ of norethindrone and ethinyl estradiol after OC alone on Day 21 of Period 1 and after OC with albiglutide on Day 21 of Period 2. | Day 21 of each period.
Predose serum levels of LH and FSH after OC alone and after OC with albiglutide. | Days 1 and 11 through 14 of each period.
Predose serum levels of progesterone after OC alone and after OC with albiglutide. | Day 21 of each period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bush M, Scott R, Watanalumlerd P, Zhi H, Lewis E. Effects of multiple doses of albiglutide on the pharmacokinetics, pharmacodynamics, and safety of digoxin, warfarin, or a low-dose oral contraceptive. Postgrad Med. 2012 Nov;124(6):55-72. doi: 10.3810/pgm.2012.11.2613. PMID 23322139
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 107032 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/107032?search=study&search_terms=107032#rs
- Available data/document: Individual Participant Data Set: 107032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register